CLINICAL TRIAL: NCT00448890
Title: Single-Blind, Randomised, Placebo-Controlled Two-Part Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Escalating Doses and Repeat Doses of GSK729327 in Healthy Volunteers
Brief Title: Evaluation of Single and Repeat Doses of GSK729327 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AM1107296
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Schizophrenia
Keywords: AMPA positive modulator, healthy volunteers
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- GSK729327 (Experimental): Dose escalation from 1.0mg to 6 mg.
  Interventions: Drug: GSK729327
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK729327 — Tablets
  Arms: GSK729327
Drug: Placebo — GSK729327 Matching placebo - Tablets
  Arms: Placebo

SUMMARY:
GSK729327 is a selective positive allosteric modulator of AMPA-type ionotropic glutamate receptors, exhibiting equivalent potency at all AMPA receptor subtypes. On the basis of preclinical studies it is expected that this compound will improve cognitive measures in schizophrenic patients with acceptable safety. This is a First Time in Human Study (FTIH) to assess the safety, tolerability, pharmacokinetics and preliminary pharmacodynamics of GSK729327 in healthy volunteers. The study will be conducted in 2 parts, with single doses being explored in Part A and multiple doses over 28 days in Part B. Part A will be a single blind, placebo controlled, single oral dose, dose-rising cross-over study in healthy male volunteers. Subjects will be randomized into two cohorts with an alternate panel design. There will be up to nine dosing sessions in total in order to investigate up to 7 different doses. The initial dose will be 0.25 mg and subsequent doses will be determined based on the pharmacokinetic and safety results from the previous dose. Part B will be a randomised, single blind, placebo-controlled, parallel group study of repeat oral dosing of GSK729327. Up to 4 cohorts of 15 (12 subjects receiving active dose and 3 subjects receiving placebo) healthy male and females of (non-childbearing potential) volunteers will be enrolled in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years inclusive.
* Part B also includes healthy female subjects of non-child bearing potential.
* A normal ECG, physical examination and laboratory screen.
* Body weight >50 kg and BMI within the range 18.5-29.9 kg/m2 inclusive.
* Signed and dated written informed consent prior to admission to the study.

Exclusion Criteria:

* Abuse of alcohol.
* A positive pre-study urine drug or alcohol screen.
* A positive pre-study HIV, Hepatitis B surface antigen or positive Hepatitis C antibody result at screening.
* History of DSM-IV alcohol and/or drug abuse or dependence.
* Consumption of grapefruit juice or grapefruit within 7 days prior to the first dose of study medication until final evaluation.
* Has received an investigational drug or has participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (which ever is longer) prior to the first dose of study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs within 4 weeks prior to the first dose of study medication until final evaluation. Where participation in study would result in donation of blood in excess of 500 ml within a 56 day period.
* History or presence of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of cholecystectomy or biliary tract disease.
* History of regular use of tobacco- or nicotine-containing products within 6 months of the start of a study.
* An unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first dose of study medication until 90 days following administration of the last dose of study medication.QTc interval > 450 ms. Or an ECG that is not suitable for QT measurements.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* The subject has a history of myocardial infarction .The subject has a resting pulse rate <55 or >100 bpm OR a systolic blood pressure >140 or <100 OR a diastolic blood pressure >90 or <60.Current or past history of symptomatic orthostatic hypotension. The subject has any laboratory abnormality that in the investigator's judgment is considered to be clinically significant (even if not outside of specified ranges).History of known or suspected seizures, including infantile febrile, unexplained significant and recent loss of consciousness or history of significant head trauma with loss of consciousness or a family history (first degree relative) of epilepsy or seizures (fits).History or presence of psychiatric disease.
* History of suicidal attempts or behavior. Subjects who cannot complete the neuropsychological test battery despite having undergone the training sessions.
* Subject has a history of sleep problems in the last 3 months.
* The subject has clinically significant abnormalities in haematology, blood chemistry, ECG, or physical examination not resolved by the screening visit. Abnormal response to photic stimulation EEG. Abnormal prolactin or TSH or free T4 or free T3 at screening/baseline.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability endpoints of AEs; EEG; ECGs; neurological assessments; vital signs and clinical laboratory values.Part A PK parameters of Cmax,AUC,t1/2,Tmax,Ae(0-t).Part B PK parameters of Cmax,Tmax,t1/2,AUC and accumulation ratio. | throughout the study

SECONDARY OUTCOMES:
Pharmacodynamic effects on Bond-Lader,Body Sway and EEG and the relationship of plasma levels of GSK729327 with pharmacodynamic parameters.Part B will also look atcognitive function,Polysomnography and LSEQ. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Berlin, State of Berlin, Germany
- GSK Investigational Site, London, United Kingdom